CLINICAL TRIAL: NCT07004959
Title: Randomised Controlled Non-inferiority Trial Comparing Vaginal Ultrasound-guided Ethanol Sclerotherapy and Laparoscopic Cystectomy for the Management of Ovarian Endometriomas
Brief Title: Non-inferiority Trial Comparing Vaginal Ultrasound-guided Ethanol Sclerotherapy and Laparoscopic Cystectomy for the Management of Ovarian Endometriomas (E-STEP)
Acronym: E-STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCAPHM20_0429
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Endometrioma
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sclerotherapy (Experimental)
  Interventions: Procedure: Vaginal ultrasound-guided ethanol sclerotherapy
- Intraperitoneal cystectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic cystectomy

INTERVENTIONS:
Procedure: Vaginal ultrasound-guided ethanol sclerotherapy — Use of an endovaginal ultrasound probe combined with a puncture guide. The technique involves locating the endometriosis cyst, echo-guided drainage via the endovaginal route, sclerotherapy (replacement of 60% of the punctured volume with 95% ethanol left in place for 10 minutes) and then reaspiration of the ethanol.
  Arms: Sclerotherapy
Procedure: Laparoscopic cystectomy — Conventional laparoscopy, with the laparoscope introduced through a 10mm incision at the umbilicus, and the laparoscopic instruments used through two or three 5mm incisions (suprapubic and right and left fossa iliaca). The surgical technique may vary according to the patient and the surgeon's preferences or habits, but must necessarily include a cystectomy (cyst wall sent for anatomopathology).
  Arms: Intraperitoneal cystectomy

SUMMARY:
Endometriosis is a disease that affects between 6 and 10% of women of childbearing age. It is defined by the presence of endometrial tissue outside the uterine cavity, most often in the ovaries or the peritoneal cavity.

The standard treatment for endometriomas is laparoscopic intraperitoneal cystectomy. This treatment has been shown to be associated with a lower rate of recurrence of painful symptoms than simple cyst drainage, and with higher pregnancy rates. Nevertheless, cystectomy can lead to a reduction in ovarian reserve due to the removal of adjacent healthy ovarian tissue, particularly when there is no cleavage plane between the ovary and the endometrioma.

Other methods have been developed to manage endometriomas while preserving the ovarian reserve. Endometrioma sclerotherapy is one of the most promising techniques for reducing the risk of recurrence while preserving the ovarian reserve. This technique involves injecting a sclerosing agent into the cystic cavity, which has been drained beforehand, in order to create an abrasion of the cystic epithelium, resulting in inflammation and fibrosis that can lead to the permanent destruction of the cyst.

The aim of the study is to conduct a single-centre randomised controlled non-inferiority trial comparing sclerotherapy and intraperitoneal cystectomy for the treatment of endometriomas.

The main hypothesis of the study is that sclerotherapy is not inferior to cystectomy in terms of reducing painful symptoms one year after the operation and that it is superior to cystectomy on one or more of the following criteria: preservation of ovarian reserve, operative complications, post-operative pain, patient acceptability/satisfaction.

The number of patients to be included will be 64, calculated to demonstrate non-inferiority between sclerotherapy and cystectomy for the primary endpoint.

DETAILED DESCRIPTION:
Endometriosis is a disease that affects between 6 and 10% of women of childbearing age. It is defined by the presence of endometrial tissue outside the uterine cavity, most often in the ovaries or the peritoneal cavity. Endometriomas are ovarian cysts whose lining is composed of ectopic endometrium and which contain a liquid resulting from the accumulation of menstrual debris. Between 17% and 44% of women with endometriosis have one or more ovarian endometriomas (i.e. between 1% and 5% of women). The clinical symptoms of endometriomas include pelvic pain (dysmenorrhoea, chronic pelvic pain or dyspareunia) and/or infertility. The standard treatment for endometriomas is laparoscopic intraperitoneal cystectomy. This treatment has been shown to be associated with a lower rate of recurrence of painful symptoms than simple cyst drainage, and with higher pregnancy rates. Nevertheless, cystectomy can lead to a reduction in ovarian reserve due to the removal of adjacent healthy ovarian tissue, particularly when there is no cleavage plane between the ovary and the endometrioma. Excessive coagulation to ensure haemostasis after cystectomy could also contribute to this reduction in ovarian reserve. Other methods have been developed to manage endometriomas while preserving the ovarian reserve: therapeutic abstention, drainage, laser or plasma energy ablation and sclerotherapy. Endometrioma sclerotherapy is one of the most promising techniques for reducing the risk of recurrence while preserving the ovarian reserve. This technique involves injecting a sclerosing agent into the cystic cavity, which has been drained beforehand, in order to create an abrasion of the cystic epithelium, resulting in inflammation and fibrosis that can lead to the permanent destruction of the cyst. This very simple technique is effective and low-risk for treating endometriomas:

* Recurrence rate between 0 and 62.5% depending on the protocol (recurrence rate after cystectomy between 6 and 67%).
* Improvement in pain in 68 to 96% of patients.
* Improvement in ovarian reserve compared with intraperitoneal cystectomy (increase in antral follicle count and AMH and higher number of oocytes harvested during subsequent in vitro fertilisation).
* Low complication rate: transient abdominal pain (1.8 - 15.3%), transient alcohol intoxication (3.8%).

Most of what is known about serotherapy comes from non-comparative prospective studies and a few randomised trials comparing sclerotherapy with either no treatment or simple drainage of the endometrioma. In addition, most studies have been conducted in the specific context of endometriomas recurring after cystectomy. To date, there is no comparative trial between sclerotherapy and intraperitoneal cystectomy (reference treatment).

We aim to conduct a single-centre randomised controlled non-inferiority trial comparing sclerotherapy and intraperitoneal cystectomy for the treatment of endometriomas.

The main hypothesis of the study is that sclerotherapy is not inferior to cystectomy in terms of reducing painful symptoms one year after the operation and that it is superior to cystectomy on one or more of the following criteria: preservation of ovarian reserve, operative complications, post-operative pain, patient acceptability/satisfaction.

The main objective is to investigate the non-inferiority of sclerotherapy of endometriomas one year after the operation in terms of reduction of painful symptoms compared with laparoscopic cystectomy. The reduction in painful symptoms was defined by the difference in the number of millimetres of VAS for pain between the preoperative consultation and the consultation one year after the operation, according to the answer to the question : " Indicate the subjective level of your endometriosis-related pain over the last 4 weeks by simply drawing a line through the line".

The secondary objectives were to compare the two techniques:

* The evolution of the 3 components of endometriosis-related pain (chronic pelvic pain, dysmenorrhoea and dyspareunia) with a VAS evaluation at 3 months and one year.
* Subjective evaluation of the evolution of treatment-related symptoms at 3 months and one year (based on self-assessment using the Clinical Global Impression Scale (CGI-S)).
* Patient satisfaction at 3 months (based on the SSQ-8 questionnaire).
* The endometrioma recurrence rate at one year (defined as the visualisation of an endometrioma with a maximum diameter greater than 3 cm on the same ovary on ultrasound or pelvic MRI one year after the operation).
* Pregnancy rate at one year for all patients (defined by at least one analysis of a quantitative plasma HCG level greater than 100 IU/ml in the year following the operation).
* The one-year pregnancy rate for patients who have expressed a desire to become pregnant within the year (defined by at least one analysis of the quantitative plasma HCG level greater than 100 IU/ml within the year following the procedure). Assessment of ovarian reserve at one year (defined by the AMH value one year after the operation and by the antral follicle count between the 2nd and 5th day of the cycle one year after the operation).
* Changes in quality of life at 3 months and one year (based on responses to the SF-36 questionnaire).
* The rate of per- and post-operative complications.
* Duration of the operation and length of post-operative hospitalisation.

The number of patients to be included will be 64, calculated to demonstrate non-inferiority between sclerotherapy and cystectomy for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 45
* Endometrioma diagnosed by endovaginal ultrasound or MRI (examinations carried out by a radiologist or gynaecologist) with a typical appearance and whose largest diameter is between 3 and 10 centimetres.
* Pain (dysmenorrhoea or chronic pelvic pain) with a VAS greater than 30 millimetres, assessed by the question "Indicate the subjective level of your endometriosis-related pain over the last 4 weeks".

Exclusion Criteria:

* Inability to speak French
* Refusal to take part in the study
* Risk factors for impaired ovarian reserve:
* Ovarian reserve already low (AMH <1,5ng/ml or Antral follicle count < 7 on the contralateral ovary
* Bilateral or multiple endometriomas (two or more endometriomas greater than 3 centimetres in diameter).
* Previous cystectomy
* Previous major peritoneal surgery causing adhesions.
* Contraindication to sclerotherapy : allergy to ethanol
* Contraindications to general anaesthesia
* Pregnant women, women in labour and nursing mothers

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-03-19 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
Difference in the number of millimetres of VAS for pain between the preoperative consultation and the consultation one year after the operation | At 12 months
  The main objective is to investigate the non-inferiority of sclerotherapy of endometriomas one year after the operation in terms of reduction of painful symptoms compared with laparoscopic cystectomy. The reduction in painful symptoms was defined by the difference in the number of millimetres of VAS for pain between the preoperative consultation and the consultation one year after the operation, according to the answer to the question : " Indicate the subjective level of your endometriosis-related pain over the last 4 weeks by simply drawing a line through the line".

SECONDARY OUTCOMES:
Pain components | At 3 and 12 months
  The evolution of the 3 components of endometriosis-related pain (chronic pelvic pain, dysmenorrhoea and dyspareunia) with a VAS evaluation at 3 months and one year.
Subjective improvement | At 3 and 12 months
  Subjective assessment of the evolution of treatment-related symptoms at 3 months and one year (based on self-assessment using the Clinical Global Impression Scale (CGI-S)).
Patient satisfaction | At 3 months
  Patient satisfaction at 3 months (according to the SSQ-8 questionnaire)
Reccurence rate | At 12 months
  The rate of recurrence of endometriomas at one year (defined as the visualisation of an endometrioma with a maximum diameter greater than 3 cm on the same ovary on ultrasound or pelvic MRI one year after the operation).
Pregnancy rate | At 12 months
  Pregnancy rate at one year for all patients (defined by at least one analysis of the quantitative plasma HCG level greater than 100 IU/ml in the year following the procedure).
Pregnancy achievement | At 12 months
  Pregnancy rate at one year for patients who have expressed a desire to become pregnant within the year (defined by at least one analysis of the quantitative plasma HCG level greater than 100 IU/ml in the year following the operation). Assessment of ovarian reserve at one year (defined by the AMH value one year after the procedure and by the antral follicle count between the 2nd and 5th day of the cycle one year after the procedure).
Quality of life | At 3 and 12 months
  Changes in quality of life at 3 months and one year (based on responses to the SF-36 questionnaire)
Complication rate | At one month
  The rate of intra- and post-operative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine NETTER, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- gynecology department APHM, Marseille, France, France

IPD SHARING:
Plan to Share IPD: No